CLINICAL TRIAL: NCT00520312
Title: Magnetic Resonance in Peripheral Arterial Disease
Brief Title: Magnetic Resonance Imaging to Identify Characteristics of Plaque Build-Up in People With Peripheral Arterial Disease
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary McDermott, Principal Investigator, Northwestern University
Other Study IDs: 1396; R01HL083064-01A2 (NIH)
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Peripheral Vascular Diseases
Keywords: Peripheral Arterial Disease; PAD; Functional Impairment; Magnetic Resonance Imaging
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, and whole blood samples are stored for future analysis
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Peripheral arterial disease (PAD) is a disease in which fatty build-up, or "plaque," accumulates in the peripheral arteries. People with PAD often experience leg pain while walking due to reduced blood flow to the legs. This study will use magnetic resonance imaging (MRI) techniques to examine how specific features of plaque build-up in the leg arteries affect walking ability, leg strength, and balance in people with PAD.

DETAILED DESCRIPTION:
Plaque build-up caused by atherosclerosis increases the risk of blood clots, heart attack, and stroke. Blockages of plaque can occur in different areas of the body. PAD, a circulatory disorder in which blockages occur in the peripheral arteries, is one manifestation of atherosclerosis. Individuals with PAD experience reduced blood flow to the legs, which may cause leg pain while walking. This study will use MRI techniques to examine how characteristics of plaque build-up in the leg arteries change over time and how this change affects function, walking ability, leg strength, and balance in people with PAD. Results from this study may be used to shape future research studies that will attempt to identify more effective treatments for people with PAD.

This study will enroll people with PAD, as well as a smaller control group of people who do not have PAD. At an initial study visit, study researchers will interview participants to collect information about their medical history, daily activity level, walking ability, and mental functioning. Blood collection and a leg MRI will occur. Also, blood flow to the legs will be measured by comparing blood pressure measurements in the arms and legs. Leg function will be measured through a series of timed walks, leg strength exercises, and muscle power exercises. Questionnaires to assess participants' medical history will be completed by each participant's primary care doctor, and study researchers will review participants' medical records. Participants with knee pain will have a knee x-ray, and participants may wear a small device called an accelerometer for 1 week to monitor physical activity levels. During the second and third study visits, occurring at one and two year follow-up, blood flow, leg function, and leg strength will be measured. If participants cannot attend either study visit, researchers may visit participants at their home or conduct an interview over the phone. Study researchers may contact participants by phone once or twice a year for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* For participants with PAD: lowest leg ankle-brachial index (ABI) less than or equal to 0.999
* For participants in the control group: lowest ABI between 1.00 to 1.30

Exclusion Criteria:

* Foot amputation, leg amputation, or gangrene
* Recent liver transplantation
* Requires oxygen on ambulation
* End stage renal disease
* Confined to a wheelchair
* Lives in a nursing home
* Low life expectancy
* Mini-Mental Status Exam (MMSE) score of less than 23 out of 30
* Communication difficulty due to language barriers
* Inability to tolerate MRI testing for any reason
* Six-minute walk performance limited primarily by pulmonary disease, legal blindness, or severe lower extremity arthritis

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ankle Brachial Index less than 1 in participants
Sampling Method: Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2007-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Functional Performance: 6-minute walk performance | Baseline, 12 months, 24 months
MRI: Mean Plaque Volume | Baseline, 24 months

SECONDARY OUTCOMES:
Four meter walking velocity (usual pace), four meter walking velocity (fastest pace), SPPB | Baseline, 12 months, 24 months
MRI: maximum plaque volume, external remodeling, mean percent lumen reduction, maximum percent lumen reduction | Baseline, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary M. McDermott, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Polonsky TS, Liu K, Tian L, Carr J, Carroll TJ, Berry J, Criqui MH, Ferrucci L, Guralnik JM, Kibbe MR, Kramer CM, Li F, Xu D, Zhao X, Yuan C, McDermott MM. High-risk plaque in the superficial femoral artery of people with peripheral artery disease: prevalence and associated clinical characteristics. Atherosclerosis. 2014 Nov;237(1):169-76. doi: 10.1016/j.atherosclerosis.2014.08.034. Epub 2014 Sep 2. PMID 25240112
- [Derived] McDermott MM, Carroll TJ, Kibbe M, Kramer CM, Liu K, Guralnik JM, Keeling AN, Criqui MH, Ferrucci L, Yuan C, Tian L, Liao Y, Berry J, Zhao L, Carr J. Proximal superficial femoral artery occlusion, collateral vessels, and walking performance in peripheral artery disease. JACC Cardiovasc Imaging. 2013 Jun;6(6):687-94. doi: 10.1016/j.jcmg.2012.10.024. Epub 2013 May 4. PMID 23647796
- [Derived] McDermott MM, Liu K, Carr J, Criqui MH, Tian L, Li D, Ferrucci L, Guralnik JM, Kramer CM, Yuan C, Kibbe M, Pearce WH, Berry J, McCarthy W, Liao Y, Xu D, Orozco J, Carroll TJ. Superficial femoral artery plaque, the ankle-brachial index, and leg symptoms in peripheral arterial disease: the walking and leg circulation study (WALCS) III. Circ Cardiovasc Imaging. 2011 May;4(3):246-52. doi: 10.1161/CIRCIMAGING.110.962183. Epub 2011 Mar 24. PMID 21436300